CLINICAL TRIAL: NCT05946330
Title: Nutritional Education Intervention in Non-Alcoholic Fatty Liver Disease -Nafld
Brief Title: Nutritional Intervention IN Nash NON-ALCOHOLIC (NAFLD).
Acronym: NUTRINAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Doutorado Enfermagem, Clinical Professor, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPRENFERMAGEM; UFPRENFERMAGEM (Other: UFParana)
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Steatohepatitis, Nonalcoholic; Steatosis; Liver Diseases; Steatohepatitis
Keywords: Adult Health, Health Education; Nutrition Literacy; Nutrition Education,; Non-Alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases; Health Education

STUDY DESIGN:
Intervention Model Description: Allocation to the intervention will be performed by simple randomization technique in a 1:1 ratio. The intervention group will receive individual nutrition education actions with nutrition consultation (in person at the beginning and at 180 days of the intervention and phone calls and text messages at 30, 60, 90, 120 and 150, 240 and 300 days of follow-up. The group The control will receive the usual care at the Outpatient Clinic. The collection of clinical, anthropometric, sociodemographic and food consumption data will be carried out during the nutrition consultations, as well as the application of the NLS-Br Nutritional Literacy questionnaire to verify literacy. During the nutrition consultation A 24-hour recall will be carried out to collect information on food consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will be followed up for one year by nutritionist intervention, on individual goals (Experimental): Patients allocated in the study will be randomized 1:1 and followed up for one (1) year, intervention group (IG) with nutritionist consultations, nutritional diagnosis and educational intervention with agreement on individual goals.
  Interventions: Behavioral: NUTRITIONAL EDUCATIONAL INTERVENTION IN FATTY LIVER DISEASE NON-ALCOHOLIC (NAFLD).
- Control Group (CG) will maintain the usual outpatient care. (Active Comparator): Patients in the Control Group (CG) will maintain the usual outpatient care.
  Interventions: Behavioral: NUTRITIONAL EDUCATIONAL INTERVENTION IN FATTY LIVER DISEASE NON-ALCOHOLIC (NAFLD).

INTERVENTIONS:
Behavioral: NUTRITIONAL EDUCATIONAL INTERVENTION IN FATTY LIVER DISEASE NON-ALCOHOLIC (NAFLD). — The intervention group will receive educational actions in individual nutrition with nutrition consultation (in person at the beginning and at 180 days of the intervention and phone calls and text messages at 30, 60, 90, 120 and 150, 240 and 300 days of follow-up

SUMMARY:
The goal of this randomized clinical trial with adults is to discuss the effectiveness of the nutritionist's educational interventions in users diagnosed with NAFLD, compared to the usual medical follow-up of users treated at the Hepatic Steatosis Ambulatory of the Complexo Hospital de Clinicas of the Federal University of Paraná (CHCUFPR) in adults diagnosed with liver disease. The sample will consist of patients routinely monitored at the Hepatic Steatosis outpatient clinic diagnosed with non-alcoholic fatty liver disease. Patients allocated in the study will be randomized 1:1 and followed up for one (1) year, intervention group (IG) with nutritionist consultations, nutritional diagnosis and educational intervention with agreement on individual goals. Patients in the Control Group (CG) will maintain the usual outpatient care. Participants will have clinical, anthropometric and sociodemographic data collected and food consumption data will be carried out during the nutrition consultations, as well as the application of the NLS-Br Nutritional Literacy questionnaire to verify literacy. During the nutrition consultation, a 24-hour recall will be carried out to collect information on food consumption. They will also be carried out as monthly telephone contacts or messages via instant messaging application, to solve the doubts of the participants and notify them of upcoming meetings, and subsequent comparison of the LN in the target population. All interventions will be recorded in specific instruments for this purpose.

Researchers will compare intervention group (IG) and Control Group (CG) and to see the effects of nutritional intervention. The expected primary outcome will be weight loss of 5% to 10% of the initial weight and the secondary outcomes will be: reduction in abdominal circumference and body mass index, and improvement in the levels of liver transaminases. Data will be analyzed with descriptive and inferential statistics.

DETAILED DESCRIPTION:
The research intends to discuss the effectiveness of the nutritionist's educational interventions in users diagnosed with NAFLD, compared to the usual medical follow-up of users treated at the Hepatic Steatosis Ambulatory of the Complexo Hospital de Clinicas of the Federal University of Paraná (CHCUFPR).

Considering:

* That NAFLD e has gained alarming proportions, affecting 25 to 30% of the world's population and its occurrence is associated with overweight, insulin resistance and metabolic syndrome;
* That the morbidity and mortality associated with NAFLD has increased significantly, along with the growth of overweight in the population, and that there is still no specific marker for the diagnosis, nor a pharmacological treatment for the disease
* That prevention and treatment are based on lifestyle changes, with the adoption of healthy eating habits, which must necessarily lead to weight loss, in order to improve the condition
* That Food and Nutrition Education (EAN) is a tool for adopting healthy eating habits;
* That the Process of Care in Nutrition (PCN) is a tool that covers the domains of action of nutritionists in their clinical practice
* That nutritional literacy, understood as the ability to process and understand nutritional information is a factor for the success of EAN;
* That EAN can be seen as a set of experiences designed to facilitate the voluntary adoption of behavioral changes related to nutrition, health and well-being; It is
* That the development of educational strategies that promote better health indicators since low LN is associated with an increase in diet-related chronic diseases.

This research is justified considering that the nutritionist's role can help reduce and improve the factors that aggravate NAFLD and improve quality of life.

RESEARCH OBJECTIVE:

MAIN GOAL

-Verify the effectiveness of the educational action of the nutritionist for NAFLD and its interference in the nutritional status of the population of users of the Hepatic Steatosis Ambulatory of the Complexo de Hospital de Clínicas of UFPR.

SPECIFIC OBJECTIVES

* To characterize the nutritional profile of users with NAFLD at the Hepatic Steatosis Outpatient Clinic of the Complexo de Hospital de Clínicas of UFPR.
* Identify the interference of educational activity in nutrition literacy
* Compare dietary, anthropometric, clinical and functional indicators after intervention;

SOCIAL RELEVANCE:

Non-alcoholic fatty liver disease (NAFLD) is currently considered an epidemic disease, with a prevalence of 10 to 24% in the general population and 57% to 74% among obese people. Its presentation and severity can vary significantly, from a simple steatosis (deposition of fatty acids without inflammation) to Non-Alcoholic Steatohepatitis (NASH) with the presence of inflammation, ballooning and liver fibrosis in its final stage. There is an association of the disease with central obesity, insulin resistance and dyslipidemia. With the increase in the incidence of overweight and Metabolic Syndrome in the general population, NAFLD has become a serious public health problem, being considered the hepatic manifestation of the Metabolic Syndrome.

In most obese individuals or with adequate body mass index (BMI), and in treatment of other comorbidities, NAFLD may be present, with or without laboratory alterations such as elevations in aminotransferase levels, and for diagnostic confirmation it is necessary to perform exams such as ultrasound, or MRI or liver biopsy.

Currently, NAFLD does not have drugs that can be used for targeted conventional treatment, as it can only be treated and alleviated by controlling metabolic disorders. Thus, the treatment of NAFLD aims to reduce insulin resistance and oxidative stress, in addition to controlling associated conditions such as obesity, diabetes mellitus, dislipidemia and also to reduce inflammation and liver fibrosis. As the clinical picture of NAFLD becomes clearer, there are also challenges to developing an effective treatment. Thus, it appears that currently there are no pharmaceutical therapies approved by the Food and Drug Administration (FDA) to treat nonalcoholic steatosis (Nonalcoholic steatohepatitis - NASH).

The improvement of the NAFLD condition necessarily involves a decrease in the mass of adipose tissue. However, it is emphatic that drastic caloric restrictions, despite leading to rapid weight loss, are not recommended due to the increased concentration of circulating fatty acids, mobilized from the adipose tissue, which can increase their influx into the liver, aggravating the condition.

Although sustained weight loss of 3% to 5% can already lead to clinically significant reductions in some cardiovascular risk factors, weight losses greater than this margin yield greater benefits. An initial goal of losing 5% to 10% of the initial weight in six months is feasible to reduce complications. For this to happen, one of the tools is diet therapy monitoring and Food and Nutrition Education (EAN).

EAN is a set of systematized strategies to encourage the culture and appreciation of food, conceived in recognition of the need to respect, but also to adjust beliefs, values, attitudes, practices and social relationships that are established around food, with a view to economic and social access to adequate food in quality and quantity, which meets the objectives of health, pleasure and social life.

Still, the strengthening of ties with the multidisciplinary team, with the inclusion of a nutritionist in the systematized diet therapy educational activity, can increase the quality of life of the population under study.

SCIENTIFIC BACKGROUND: In the world, malnutrition in all its forms, including malnutrition, obesity and other dietary risks, for the development of chronic non-communicable diseases (NCDs), corresponds to 19% of the causes of illnesses and premature deaths in everyone. Among the NCDs related to malnutrition, non-alcoholic fatty liver disease (NAFLD) stands out, a syndrome that occurs in non-alcoholic patients, but who present liver damage histologically indistinguishable from alcoholic steatohepatitis.

CASUISTRY Nutritional intervention, when followed correctly, is effective in treating NAFLD in patients who achieve a minimum weight loss of 5% of their baseline body weight after 6 months of dietary therapy. Important alterations in the parameters of insulin resistance and metabolic syndrome are observed in these patients. Even an average reduction of only 2% of the initial body weight (non-adherent group) led to a decrease in some anthropometric parameters, such as BMI and waist circumference, when compared with baseline values. However, patients who lost at least 5% of their initial weight (adherent group) showed more pronounced reductions in these parameters, in addition to improvements in waist-hip ratio, glucose, insulin, HDL-C and LDL-C, alterations not observed in patients non-adherent.

RESEARCH MATERIAL:

For data collection, a form with clinical, dietary and socioeconomic data prepared by the researchers will be used. For the analysis of food intake, a 24-hour recall will be used and the assessment of Nutritional Literacy will be measured using the Nutritional Literacy Scale - NLS - Brazilian version.

PROPOSED METHOD:

Randomized controlled clinical trial with division into two groups (GI and CG) matched 1 to 1. Essentially, it is a study in which participants already seen at the Hepatic Steatosis Outpatient Clinic will be invited to participate and will be randomly allocated (participants are randomized) to receive one or more interventions. Clinical trial results can be directly incorporated into everyday clinical practice. Allocation to the intervention will be performed by simple randomization technique in a 1:1 ratio.

The intervention group will receive individual nutrition education actions with nutrition consultation (in person at the beginning and at 180 days of the intervention and phone calls and text messages at 30, 60, 90, 120 and 150, 240 and 300 days of follow-up. The group The control will receive the usual care at the Outpatient Clinic. The collection of clinical, anthropometric, sociodemographic and food consumption data will be carried out during the nutrition consultations, as well as the application of the NLS-Br Nutritional Literacy questionnaire to verify literacy. During the nutrition consultation A 24-hour recall will be carried out to collect information on food consumption.

They will also be carried out as monthly telephone contacts or messages via instant messaging application, to solve the doubts of the participants and notify them of upcoming meetings, and subsequent comparison of the LN in the target population. All interventions will be recorded in specific instruments for this purpose

EXPECTED OUTCOME It is expected that patients assisted by the nutritionist will have an improvement in the prognosis of non-alcoholic fatty liver disease (NAFLD), reduction in body weight and centripetal adipose mass, modification of lifestyle and increase in nutritional literacy.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory users with a diagnosis of NAFLD in the medical record will be included. For the purposes of eligibility of the patient under study, users must not be significant alcoholics and this questioning, self-reported, is provided for in the nutritionist's consultation protocol. Alcohol consumption is considered significant if defined as > 21 drinks per week in men and > 14 drinks per week in women in a two-year period prior to baseline liver histology.

Exclusion Criteria:

People who are not able to answer the nutritional literacy questionnaire with the help of the researcher will not be included in the research or who, during the research, show accumulation of hepatic fat due to secondary causes, such as the use of steatogenic drugs or hereditary diseases, as well as patients who report frequent alcohol intake. Patients with positive serology for hepatitis B and C, HIV, as well as patients with disabsorptive diseases (Chron's Disease, Celiac Disease), with chronic kidney diseases, who are on the waiting list for bariatric surgery, pregnant and lactating women will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss of 5% to 10% of body weight, decrease in waist circumference (WC) | changes at 180 and 360 days.
  The primary clinical outcomes expected for this study are weight loss of 5% to 10% of body weight, decrease in waist circumference (WC), as well as changes in dietary intake pattern, laboratory and anthropometric changes at 180 and 360 days.

SECONDARY OUTCOMES:
Cessation of the progression of NAFLD | changes in 180 and 360 days
  Cessation of the progression of NAFLD, through liver enzymes, improvement in the prognosis of cure of NAFLD, continued slimming, improvement in consumption pattern, with comparison of three food recalls, improvement in self-reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Mantovani, Dr, Principal Investigator — Universidade Federal do Paraná; Maria E Schieferdecker, Dr, Study Chair — Universidade Federal do Paraná
Locations (1):
- Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
In the Informed Consent Form (TCLE), signed by the participants, I affirm that the collected data will not be shared with other studies.

REFERENCES:
- See also: The Brazilian Registry of Clinical Trials (ReBEC) is a free access virtual platform for recording experimental and non-experimental studies carried out on human beings and conducted in Brazilian territory, by Brazilian and foreign researchers. — https://ensaiosclinicos.gov.br/welcome